CLINICAL TRIAL: NCT05839795
Title: Evaluation of Musculoskeletal System in Caregivers of Rehabilitation Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Halime Arikan, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 83116987-271
Record Dates: First submitted 2023-04-18; First posted 2023-05-03 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2023-09

CONDITIONS: Caregiver Burden; Stroke; Cerebral Palsy; Neurologic Disorder; Pediatric Disorder; Orthopedic Disorder
Keywords: Pain; Caregiver; Low back; Neck; Musculoskeletal system
MeSH Terms: conditions — Caregiver Burden; Stroke; Cerebral Palsy; Nervous System Diseases; Musculoskeletal Diseases; Pain | interventions — Outcome Assessment, Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Caregivers of Rehabilitation Patients (Other): Caregivers of rehabilitation patients, such as those with neurological, pediatric, and orthopedic disorders
  Interventions: Other: Assessment study

INTERVENTIONS:
Other: Assessment study — Evaluation of musculoskeletal-related pain, posture, spine function, lumbar and neck regions, musculoskeletal disorder, fatigue, and quality of life

SUMMARY:
In this study, musculoskeletal-related pain, posture, spine function, the condition of the low back and neck regions, musculoskeletal system disorders, fatigue, and quality of life will be examined in caregivers of rehabilitation patients.

DETAILED DESCRIPTION:
There are studies examining musculoskeletal disorders, physical demands and care activities of unpaid caregivers, musculoskeletal pain and related factors in unpaid caregivers of individuals with stroke, the effect of the functional status of stroke individuals on caregiver pain, musculoskeletal pain and related factors in mothers of children with cerebral palsy, musculoskeletal symptoms in caregivers of individuals with stroke, the prevalence of musculoskeletal disorders in caregivers of individuals with disabilities in a rehabilitation center, and the prevalence and characteristics of low back pain in caregivers of individuals with stroke in the literature. However, no study was found in which the musculoskeletal system was comprehensively evaluated in the caregivers of rehabilitation patients and the musculoskeletal system characteristics were compared in the caregivers of individuals with cerebral palsy and stroke. Therefore, musculoskeletal-related pain, posture, spine function, the condition of the low back and neck regions, musculoskeletal system disorders, fatigue, and quality of life will be examined in caregivers of rehabilitation patients in this study.

ELIGIBILITY:
Inclusion Criteria:

* The caregiver of the rehabilitation patient,
* Can speak, read, write Turkish,
* Over 18 years old.

Exclusion Criteria:

* Pregnant,
* Can't speak, read or write Turkish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2025-01-04 (Actual)

PRIMARY OUTCOMES:
Musculoskeletal-related pain | through study completion, an average of 6 month
  Musculoskeletal related pain will be evaluated with the Numeric Pain Rating Scale. The scale starts with 0 (no pain) and ends with 10 (unbearable pain). A score is obtained by measuring the value marked on the scale in the evaluation.
Posture | through study completion, an average of 6 month
  The New York Posture Evaluation Scale will be used to evaluate the posture of individuals. The scale, which examines the alignment of the body parts in the anatomical position, divides the body into 13 parts and provides the opportunity to evaluate from two different directions (anterior, lateral). Scoring is done in the form of "1", "3", "5". 1 point means severely impaired, 3 points means moderately impaired, and 5 points means proper posture. The total score ranges from 13-65. A high score means good posture.
Spine function | through study completion, an average of 6 month
  The Spine Functions Index is a 25-item scale developed to examine the effect of spine-related symptoms on functionality. Each question is scored as "0", "0.5", and "1". The total score is calculated as a percentage, and a score closer to 100 indicates normal spine functions.
Lumbar impairment | through study completion, an average of 6 month
  The Modified Oswestry Disability Index includes 10 questions about pain intensity, personal care, weight lifting, walking, sitting, standing, sleeping, social life, travel and change in pain over time, each question has 6 options. The individual is asked to choose the one that best describes his/her situation from the options between 0 and 5 points in each question. The highest score is 50 points. An increase in the score indicates an increase in functional limitation, while a decrease in the score indicates an increase in functional level.
Neck impairment | through study completion, an average of 6 month
  The Bournemouth Neck Questionnaire will be used to evaluate individuals in terms of neck pain severity, participation in family and social life, depression, anxiety, kinesiophobia, and ability to cope with pain. It consists of 7 questions in total and each question is scored between 0 and 10. A higher score means more impairment.
Musculoskeletal disorder | through study completion, an average of 6 month
  To assess musculoskeletal discomfort, the Cornell Musculoskeletal Discomfort Questionnaire will be used. The Cornell Musculoskeletal Discomfort Questionnaire collects information on the severity of discomfort as well as the effects of the condition for specific regions of the human body. The survey is also a one-page chart that combines the frequency and intensity of musculoskeletal pain and complaints with work-related impairments for 20 body regions.
Fatigue | through study completion, an average of 6 month
  The fatigue of caregivers will be evaluated with the Fatigue Severity Scale. The person indicates how much he or she agrees with each item by choosing numbers from 1 to 7. 1 means completely disagree, 7 means completely agree. The score range of the scale, which consists of 9 questions in total, is 9-63. A score of 36 or higher indicates severe fatigue.
Quality of life of caregivers | through study completion, an average of 6 month
  Short Form-36 is one of the most common generic measures used to measure quality of life. This scale examines 8 dimensions of health with 36 items, such as physical function, role limitations (due to physical and emotional problems), social function, mental health, vitality (energy), pain and general perception of health. A high score indicates a low quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Researchers involved in the study will have individual data.